CLINICAL TRIAL: NCT03279809
Title: The Effect of Aspirin on Patency of Metal Stent in Malignant Distal Bile Duct Obstruction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: One grade 4 adverse event (AE) and common (47.2%) grade 3 AEs
Sponsor: Woo Hyun Paik (Other)
Responsible Party: Sponsor-Investigator, Woo Hyun Paik, Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-1707-161-874
Record Dates: First submitted 2017-09-05; First posted 2017-09-12 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Biliary Stasis, Extrahepatic
MeSH Terms: conditions — Cholestasis, Extrahepatic | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention : aspirin medication Case with aspirin medication for 6 months after stenting
  Interventions: Drug: Aspirin
- Control (Placebo Comparator): Control : placebo medication Case with placebo medication for 6 months after stenting
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — Aspirin medication (100mg daily) after biliary stent insertion for malignant obstruction
  Other Names: Aspirin 100 mg
  Arms: Intervention
Drug: Placebo — Case with placebo medication for 6 months after stenting
  Other Names: Placebo drug of aspirin
  Arms: Control

SUMMARY:
The aim of this study is to determine whether administration of aspirin can help maintain the patency of metallic stents for distal malignant common bile duct obstruction. Metal stents are mainly used for malignant biliary obstruction if the surgical treatment is not considered and its maintenance period has been reported to be about 8 months. This study will be prospectively conducted as a randomized controlled study with aspirin treated patients who received metal stents in patients over 20 years who were confirmed malignant distal biliary obstruction. The primary endpoint is the incidence of stent dysfunction in both groups for 6 months after the procedure. The secondary endpoints included duration of metallic stent patency, incidence of further procedures, and adverse events related with aspirin.

DETAILED DESCRIPTION:
Background -Endoscopic drainage is the first choice for bile drainage in patients with malignant distal biliary obstruction. Metal stents are mainly used for malignant biliary obstruction if the surgical treatment is not considered. Metal stents have proven superior in many clinical aspects over plastic stents. Nonetheless, the maintenance period of the metallic stent patency has been reported to be around 8 months, and it is often necessary to undergo further procedure due to dysfunction of stents. Recently, it has been reported that the duration of the metallic stent patency in patients with aspirin is prolonged. Since the previous study was a retrospective study, this study will be prospectively conducted as a randomized controlled study with aspirin treated patients who received metal stents in patients over 20 years who were confirmed malignant distal biliary obstruction. The incidence of stent dysfunction in both groups for 6 months after the procedure will be compared. Stent dysfunction is defined as any case which further procedure is required due to jaundice or cholangitis after stent insertion.

Study aim

-The aim of this study is to determine whether administration of aspirin can help maintain the patency of metallic stents for distal malignant common bile duct obstruction.

Data analysis

* Blinding will remain in place until the statistician codes the statistical analyses of the primary and secondary outcomes. The statistical analyses will be done using the full analysis set according to the intention-to-treat principle, meaning all the randomized patients will be analyzed in their allocated groups regardless of any protocol violations or early treatment discontinuations. The outcomes through a per-protocol analysis set that will consider only the subjects who followed the protocol effectively will be analyzed.
* The rate of stent dysfunction will be compared using Pearson's chi-squared test with Fisher's exact test and calculated the odds ratio of the event. The secondary outcomes (i.e., the duration of stent patency, the rate of reintervention, and the adverse events related to aspirin administration) will be analyzed using Pearson's chi-squared test with Fisher's exact test, Student's t-test, and Kaplan-Meier curves stratified by drug and the hazard ratios between two groups using the Cox proportional hazards. The further affecting factors for stent dysfunction will be assessed by univariable and multivariable logistic regression analysis.
* In the initial plan, it was decided not to perform interim analysis, but it was confirmed that more adverse events occurred than expected in the process of conducting the study. Therefore, the interim analysis was performed with the data up to May 2020, and determine whether to continue the study by measuring the benefits and losses obtained from aspirin.

ELIGIBILITY:
Inclusion Criteria:

* Malignant distal bile duct obstruction
* Over 20 years old
* Techinical success of endoscopic retrograde biliary drainage with metalic stent

Exclusion Criteria:

* Patient's denial
* Previous Aspirin use
* Aspirin allergy
* Contraindication for aspirin
* Life expectancy < 6mo
* Gastroduodenal ulcer
* History of substance abuse
* Participation in a clinical trial within the past 30 days

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2020-09-05 (Actual); Study Completion 2020-09-05 (Actual)

PRIMARY OUTCOMES:
Incidence of stent dysfunction | 6 months after biliary metalic stent
  Dysfunction after 6 months from stenting

SECONDARY OUTCOMES:
Duration of metalic stent patency | 6 months after biliary metalic stent
  Duration from insertion time to metallic stent dysfunction time
Incidence of further procedures | 6 months after biliary metalic stent
  Incidence of further procedures needed for biliary drainage
Adverse events related with aspirin | 6 months after biliary metalic stent
  Adverse events which clearly related with aspirin admistration including bleeding event

CONTACTS AND LOCATIONS:
Overall Officials: Woo Hyun Paik, MD, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Choi JH, Paik WH, You MS, Lee KJ, Choi YH, Shin BS, Lee SH, Ryu JK, Kim YT. Aspirin for metal stent in malignant distal common bile duct obstruction (AIMS): study protocol for a multicenter randomized controlled trial. Trials. 2020 Jan 30;21(1):120. doi: 10.1186/s13063-020-4083-z. PMID 32000828